CLINICAL TRIAL: NCT04157010
Title: Prospective, Single-centre, Open-Label, Randomised, Pilot Study Assessing the Changes in Expression of Janus Kinase/Signal Transducers and Activators of Transcription (JAK-STAT) and Speed & Depth of Remission Induced by Tocilizumab & Methotrexate Combination and Tocilizumab Monotherapy in Patients With Early Rheumatoid Arthritis
Brief Title: Tocilizumab REMission in Early RA
Acronym: TREMERA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Principal Investigator, Dr Maya Buch, Chief Investigator, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RR11/9965; 2011-004017-17 (EudraCT Number); 14383 (Other: UKCRN)
Record Dates: First submitted 2014-04-15; First posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TCZ monotherapy (Experimental): Tocilizumab (TCZ) monotherapy 8mg/kg 4-weekly for a total of 48 weeks.
  Interventions: Drug: Tocilizumab
- TCZ+MTX combination therapy (Experimental): Tocilizumab (TCZ) and methotrexate (MTX) combination therapy 8mg/kg 4-weekly for a total of 48 weeks.
  Interventions: Drug: Tocilizumab; Drug: Methotrexate

INTERVENTIONS:
Drug: Tocilizumab
Drug: Methotrexate
  Arms: TCZ+MTX combination therapy

SUMMARY:
The TREMERA study focuses on patients with newly diagnosed, untreated, rheumatoid arthritis (RA). Recent international treatment recommendations emphasise the need to diagnose RA early and start treatment immediately (this being associated with better response rates); and to aim for the goal of remission i.e. the absence of signs and symptoms of active inflammatory disease activity which is associated with better outcomes for the patient. Remission is more achievable with significant treatment advances that have been made in the form of highly effective biologic therapies. Tocilizumab (TCZ) is a newly introduced biologic drug that is used in established RA. The TREMERA study primarily aims to investigate the biological changes seen in blood and tissue following TCZ therapy this will contribute to a better understanding of how the drug works as well as disease processes; and will also identify whether administering a biologic drug such as TCZ can also switch off immunological parameters associated with a disrupted immune system of RA. The study will assess the effectiveness of TCZ given on its own or in combination with methotrexate (MTX; a standard therapy usually given with biologic treatments)in patients with early onset RA to determine the proportion that achieve remission. This study also aims to find out how quickly remission can be achieved with TCZ and the depth of remission achieved. This will be done using usual clinical assessment but also imaging such as ultrasound and magnetic resonance imaging (MRI) which can detect inflammation not apparent on clinical assessment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of rheumatoid arthritis (2010 ACR/EULAR RA classification criteria)
* Symptom duration ≤12months
* No previous disease modifying antirheumatic drug (DMARD) therapy
* Active RA at baseline (defined as: DAS28 ≥ 3.2)
* Active hand and/or wrist joint evaluable by US and MRI (with no planned surgery during the study period)
* Patients without any contraindication to MRI

Exclusion Criteria:

* Patients unwilling or unable to receive MTX for the duration of the study.
* Patients with inflammatory joint disease of different origin, mixed connective tissue disease, Reiter's syndrome, psoriatic arthritis, systemic lupus erythematosis, or any arthritis with onset prior to 16 years of age.
* Suspicion of diagnosis of tuberculosis (TB): positive quantiferon +/abnormal chest x-ray, as per clinician judgement. Prior history of TB with confirmed full chemotherapy +/latent TB adequately treated may be included as per physician's discretion.
* Intramuscular, oral or intraarticular (of non-target joint) corticosteroid within 28 days of the screening visit; intra-articular steroid of the chosen target joint within 12 weeks of screening.
* Patients with serious infections within 3 month of enrolment (screening) or persistent infections.
* Patients at significant risk of infection (e.g. leg ulceration, indwelling urinary catheter, septic joint within 1 year (or ever if prosthetic joint still in situ).
* Known positive serology for hepatitis B or C, or HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-05; Primary Completion 2016-03-29 (Actual); Study Completion 2016-03-29 (Actual)

PRIMARY OUTCOMES:
Evaluate change in expression of JAK 1 and 3 (as well as STAT and p38 MAPK). | To week 60
  Changes up to week 60

SECONDARY OUTCOMES:
Reduction in inflammation in each treatment arm using ultrasound | To week 48
  Establish reduction in inflammation in each treatment arm using ultrasound using grey scale power doppler
Disease Activity Score (DAS): DAS28/44 remission | To week 48
  Proportion of patients achieving DAS28/44 remission
Questionnaires and research tools | Week 48
  Using tools including DAS28/44, SDAI, CDAI
Health Assessment Questionniaire (HAQ) scores | To week 48
  The change from baseline in HAQ scores.
VAS scores questionnaire | To week 48
  The change in VAS scores for pain, disease activity
Rheumatoid Arthritis Quality of Life (RAQoL) questionnaire | To week 48
  The change in RAQoL from baseline
Bone densitometry | Week 48.
  Bone densitometry scan of hands, spine, femoral neck
Sharp score on plain radiographs | Week 48.
  Change in modified Sharp score on plain radiographs

OTHER OUTCOMES:
MRI sub-study (separately consented) - optional | To week 48
  Establish if reduction in RA MRI Scoring system (RAMRIS) synovitis score
Cardiovascular sub-study (separately consented) - optional | To week 48
  Change in cardiovascular measures on cardiac MRI and serum biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Dr Maya H Buch, Principal Investigator — University of Leeds
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire, United Kingdom